CLINICAL TRIAL: NCT01255657
Title: A Phase 1 Study of ABT-806 in Subjects With Advanced Solid Tumor Types Likely to Either Overexpress Wild-Type Epidermal Growth Factor Receptor (EGFR) or to Express Variant III Mutant EGFR
Brief Title: A Study of ABT-806 in Subjects With Advanced Solid Tumor Types
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AbbVie (prior sponsor, Abbott) (Industry)
Responsible Party: Sponsor
Organization: AbbVie (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M11-847
Record Dates: First submitted 2010-11-22; First posted 2010-12-07 (Estimated); Last update posted 2017-11-21 (Actual); Status verified 2013-01

CONDITIONS: Advanced Solid Tumors
MeSH Terms: interventions — depatuxizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ABT-806 Arm (Experimental)
  Interventions: Drug: ABT-806

INTERVENTIONS:
Drug: ABT-806 — ABT-806 will be administered by intravenous infusion.

SUMMARY:
This is an open-label study designed to determine the recommended Phase 2 dose (RPTD) and evaluate the safety and pharmacokinetics of ABT-806 in subjects with advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Subject has a solid tumor of a type known to either over-express wild-type EGFR or to express variant III mutant EGFR (e.g., head and neck squamous cell carcinoma, non small cell lung cancer (NSCLC), colorectal carcinoma) or a tumor known to be EGFR positive.
* Subject must have disease that is not amenable to surgical resection or other approved therapeutic options with curative intent.
* Subject has an Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 to 2.
* Subject must have measurable disease per Response Evaluation Criteria In Solid Tumors (RECIST) version 1.1.
* Inclusion criteria for Expand Safety Cohort B - subject has histologically confirmed supratentorial glioblastoma multiforme (GBM) .

Exclusion Criteria:

* Subject has uncontrolled metastases to the central nervous system. Subjects with brain metastases are eligible provided they have shown clinical and radiographic stable disease for at least 1 month after definitive therapy. Subjects with glioblastoma multiforme (GBM) are excluded from the dose escalation portion of the study, but may be enrolled in the expanded safety cohort.
* Subject has received anticancer therapy including chemotherapy, immunotherapy, radiotherapy, hormonal, biologic, or any investigational therapy within a period of 21 days prior to the first dose of ABT-806.
* Subject has had any adjustments of an ongoing steroid medication during the 14 days prior to the first dose of ABT-806.
* Subject has received a prior EGFR-directed monoclonal antibody within a period of 4 weeks prior to the first dose of ABT-806.
* Subject has unresolved clinically significant toxicities from prior anticancer therapy, defined as any Common Terminology Criteria for Adverse Events (CTCAE) Grade 2 or higher.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2010-11; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Safety (Number of subjects with adverse events and/or dose-limiting toxicities) | At each treatment visit (weekly for first 4 weeks and then at least every 4 weeks through end of treatment)
  Evaluation of vital signs, clinical lab testing and adverse event monitoring (every other week), physical exam (every 4 weeks) and ECG (periodic)
Pharmacokinetic profile (assay for ABT-806) Dose Escalation Cohort | Week 1, 2, 3, 5, 7, 8, 9, 11, 13, 15, 19, 23 and Final Visit
  Assay for ABT-806
Pharmacokinetic profile (assay for ABT-806) Expanded Safety Cohort | Week 1, 3, 5, 7, 11, 13, 15, 19, 23 and 30 Day Follow-up
  Assay for ABT-806

SECONDARY OUTCOMES:
Pharmacokinetic profile (assay for Anti-drug Antibody) Dose Escalation Cohort | Week 1, 3, 7, 11, 15, 19, 23 and Final Visit
  Assay for Anti-drug antibody against ABT-806
QT assessment | Week 1, 7, 13, and 30 day follow-up visit
  Triplicate ECGs
Infusion rate evaluation (Expanded Safety Cohort) | Every other week
  Two infusion times explored
Pharmacokinetic profile (assay for Anti-drug Antibody) Expanded Safety Cohort | Week 1, 3, 7, 11, 15, 19, 23 and 30 Day Follow-up
  Assay for Anti-drug antibody against ABT-806

CONTACTS AND LOCATIONS:
Overall Officials: Kyle D. Holen, MD, Study Director — AbbVie
Locations (3):
- United States (3):
  - Site Reference ID/Investigator# 54056, Baltimore, Maryland
  - Site Reference ID/Investigator# 41931, Boston, Massachusetts
  - Site Reference ID/Investigator# 43422, Tacoma, Washington

REFERENCES:
- [Result] Sharma S, Mittapalli RK, Holen KD, Xiong H. Population Pharmacokinetics of ABT-806, an Investigational Anti-Epidermal Growth Factor Receptor (EGFR) Monoclonal Antibody, in Advanced Solid Tumor Types Likely to Either Over-Express Wild-Type EGFR or Express Variant III Mutant EGFR. Clin Pharmacokinet. 2015 Oct;54(10):1071-81. doi: 10.1007/s40262-015-0258-2. PMID 25761639